CLINICAL TRIAL: NCT01058668
Title: A Double-Blind, Placebo-Controlled, Evaluation of the Safety and Efficacy of Cariprazine in Patients With Acute Mania Associated With Bipolar I Disorder
Brief Title: Safety and Efficacy of Cariprazine for Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-33
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Mania; Bipolar I Disorder
Keywords: Acute Mania; Bipolar I Disorder
MeSH Terms: conditions — Mania | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cariprazine (3-6 mg/day) (Experimental): Cariprazine 3 milligrams (mg) - 6 mg capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Cariprazine
- Cariprazine (6-12 mg/day) (Experimental): Cariprazine 6 mg - 12 mg capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Placebo dose-matching cariprazine capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Patients who meet eligibility criteria will be administered a once daily oral dose of cariprazine for three weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Arms: Cariprazine (3-6 mg/day); Cariprazine (6-12 mg/day)
Drug: Placebo — Patients who meet eligibility criteria will be administered a once daily oral dose of placebo for three weeks.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of cariprazine monotherapy versus placebo for the treatment of acute manic or mixed episodes associated with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed consent prior to any study specific procedures
* Patients currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for bipolar I disorder, as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID) manic or mixed type with or without psychotic symptoms
* Voluntarily hospitalized for current manic episode
* Patients with normal physical examination, laboratory, vital signs,and/ or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of an axis I disorder other than bipolar I disorder that was the primary focus of treatment within the previous six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Diaz, MD, Study Director — Forest Laboratories
Locations (66):
- United States (23):
  - Forest Investigative Site 018, Little Rock, Arkansas
  - Forest Investigative Site 012, Cerritos, California
  - Forest Investigative Site 010, Costa Mesa, California
  - Forest Investigative Site 005, Oceanside, California
  - Forest Investigative Site 023, San Diego, California
  - Forest Investigative Site 017, San Diego, California
  - Forest Investigative Site 024, Santa Ana, California
  - Forest Investigative Site 016, New Britain, Connecticut
  - Forest Investigative Site 007, Washington D.C., District of Columbia
  - Forest Investigative Site 002, Kissimmee, Florida
  - Forest Investigative Site 003, Orlando, Florida
  - Forest Investigative Site 026, Atlanta, Georgia
  - Forest Investigative Site 013, Honolulu, Hawaii
  - Forest Investigative Site 011, Hoffman Estates, Illinois
  - Forest Investigative Site 021, Greenwood, Indiana
  - Forest Investigative Site 001, Shreveport, Louisiana
  - Forest Investigative Site 006, Rockville, Maryland
  - Forest Investigative Site 025, St Louis, Missouri
  - Forest Investigative Site 008, Cedarhurst, New York
  - Forest Investigative Site 019, Philadelphia, Pennsylvania
  - Forest Investigative Site 015, Memphis, Tennessee
  - Forest Investigative Site 004, Irving, Texas
  - Forest Investigative Site 014, Bothell, Washington
- Croatia (4):
  - Forest Investigative Site 607, Rijeka
  - Forest Investigative Site 602, Zagreb
  - Forest Investigative Site 605, Zagreb
  - Forest Investigative Site 606, Zagreb
- Romania (11):
  - Forest Investigative Site 210, Craiova, Dolj
  - Forest Investigative Site 204, Târgovişte, Dâmbovița County
  - Forest Investigative Site 211, Timișoara, Timiș County
  - Forest Investigative Site 212, Focşani, Vrancea
  - Forest Investigative Site 209, Arad
  - Forest Investigative Site 203, Bucharest
  - Forest Investigative Site 205, Bucharest
  - Forest Investigative Site 206, Bucharest
  - Forest Investigative Site 208, Bucharest
  - Forest Investigative Site 202, Constanța
  - Forest Investigative Site 201, Craiova
- Russia (9):
  - Forest Investigative Site 501, Lipetsk
  - Forest Investigative Site 503, Moscow
  - Forest Investigative Site 507, Moscow
  - Forest Investigative Site 510, Moscow
  - Forest Investigative Site 506, Saint Petersburg
  - Forest Investigative Site 508, Saint Petersburg
  - Forest Investigative Site 509, Samara
  - Forest Investigative Site 504, Saratov
  - Forest Investigative Site 502, Smolensk
- Serbia (5):
  - Forest Investigative Site 403, Belgrade
  - Forest Investigative Site 404, Belgrade
  - Forest Investigative Site 405, Belgrade
  - Forest Investigative Site 402, Kragujevac
  - Forest Investigative Site 401, Senta
- Ukraine (14):
  - Forest Investigative Site 308, Dnipropetrovsk
  - Forest Investigative Site 315, Dnipropetrovsk
  - Forest Investigative Site 301, Donetsk
  - Forest Investigative Site 307, Kharkiv
  - Forest Investigative Site 310, Kharkiv
  - Forest Investigative Site 304, Kyiv
  - Forest Investigative Site 305, Kyiv
  - Forest Investigative Site 303, Kyiv
  - Forest Investigative Site 309, Kyiv
  - Forest Investigative Site 312, Kyiv
  - Forest Investigative Site 306, Luhansk
  - Forest Investigative Site 311, Lviv
  - Forest Investigative Site 302, Odesa
  - Forest Investigative Site 314, Poltava

REFERENCES:
- [Derived] McIntyre RS, Masand PS, Earley W, Patel M. Cariprazine for the treatment of bipolar mania with mixed features: A post hoc pooled analysis of 3 trials. J Affect Disord. 2019 Oct 1;257:600-606. doi: 10.1016/j.jad.2019.07.020. Epub 2019 Jul 5. PMID 31344528
- [Derived] Earley W, Durgam S, Lu K, Ruth A, Nemeth G, Laszlovszky I, Yatham LN. Clinically relevant response and remission outcomes in cariprazine-treated patients with bipolar I disorder. J Affect Disord. 2018 Jan 15;226:239-244. doi: 10.1016/j.jad.2017.09.040. Epub 2017 Sep 25. PMID 29017067
- [Derived] Calabrese JR, Keck PE Jr, Starace A, Lu K, Ruth A, Laszlovszky I, Nemeth G, Durgam S. Efficacy and safety of low- and high-dose cariprazine in acute and mixed mania associated with bipolar I disorder: a double-blind, placebo-controlled study. J Clin Psychiatry. 2015 Mar;76(3):284-92. doi: 10.4088/JCP.14m09081. PMID 25562205

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment Phase
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-12 mg/Day)
Started | 161 | 167 | 169
Completed | 122 | 129 | 119
Not Completed | 39 | 38 | 50
Not completed — Adverse Event | 8 | 15 | 25
Not completed — Insufficient Therapeutic Response | 15 | 2 | 5
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Withdrawal of Consent | 14 | 18 | 17
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Other Unspecified | 1 | 1 | 0
Period: Safety Follow-up
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-12 mg/Day)
Started | 144 (Not all participants entered the Safety-Follow-up) | 146 | 148
Completed | 139 | 146 | 141
Not Completed | 5 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-12 mg/Day) | Total
Number analyzed (Participants) | 161 | 167 | 169 | 497
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (11.4) | 43.1 (12.2) | 41.2 (11.3) | 41.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 77 | 84 | 233
  Male | 89 | 90 | 85 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 4 | 24
  Not Hispanic or Latino | 151 | 157 | 165 | 473
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 114 | 117 | 114 | 345
  Black/African American | 44 | 44 | 51 | 139
  Asian | 1 | 3 | 1 | 5
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 0 | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 81.70 (15.96) | 82.42 (16.22) | 81.49 (16.78) | 81.87 (16.30)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.93 (9.88) | 170.99 (9.15) | 170.25 (9.36) | 170.72 (9.45)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/meter(m)^2] | 27.99 (5.15) | 28.22 (5.29) | 28.04 (4.92) | 28.08 (5.12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score at Week 3
Description: The YMRS is an 11-item scale that assesses manic symptoms based on the participant's perception of his or her condition over the previous 48 hours, as well as the physician's clinical observations during the interview. The 11-items are elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, rate and amount of speech, language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight. The severity of the abnormality for 7-items are rated on a five-point scale (0-4) and 4-items on a nine-point scale (0-8). The individual scores are summed for a total possible score of 0 (best) to 60 (worst). A negative change from Baseline indicates improvement. Analysis is a mixed model for repeated measurements (MMRM) using observed cases, with treatment group, pooled study center, visit, treatment group-by-visit interaction as factors, baseline value and baseline-by-visit interaction as covariates and an unstructured covariance matrix.
Time Frame: Baseline, Week 3
Population: Intent-to-treat Population included all participants who received at least 1 dose of study drug and who had at least 1 post-baseline YMRS assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-12 mg/Day)
Number analyzed (Participants) | 160 | 165 | 167
score on a scale | -12.5 (0.8) | -18.6 (0.8) | -18.5 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine (3-6 mg/Day); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -6.1, 95% CI 2-sided [-8.4 to -3.8] — cariprazine (3-6 mg/day) - placebo
Statistical Analysis 2: Comparison: Placebo vs Cariprazine (6-12 mg/Day); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -5.9, 95% CI 2-sided [-8.2 to -3.6] — cariprazine (6-12 mg/day) - placebo

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Total Score at Week 3
Description: The CGI-S measures the investigator's assessment of overall severity of the participant's illness compared with the severity of illness in other patients the physician has observed using a 7-point scale (1=Normal, not ill at all to 7= Among the most extremely ill participants). A negative change from Baseline indicates improvement. Analysis is based on a MMRM using the observed cases data, with treatment group, pooled study center, visit, treatment group-by-visit interaction as factors, baseline value and baseline-by-visit interaction as covariates and an unstructured covariance matrix.
Time Frame: Baseline, Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-12 mg/Day)
Number analyzed (Participants) | 160 | 165 | 167
score on a scale | -1.3 (0.1) | -1.9 (0.1) | -1.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine (3-6 mg/Day); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.4] — cariprazine (3-6 mg/day) - placebo
Statistical Analysis 2: Comparison: Placebo vs Cariprazine (6-12 mg/Day); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3] — cariprazine (6-12 mg/day) - placebo

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose (Up to 51 days)
Description: Safety Population included all participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-12 mg/Day)
Serious Adverse Events (participants affected / at risk) | 5/161 | 9/167 | 5/169
Other Adverse Events (participants affected / at risk) | 63/161 | 89/167 | 90/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Cariprazine (3-6 mg/Day) (N=167) | Cariprazine (6-12 mg/Day) (N=169)
Mania (Psychiatric disorders) | 3 | 3 | 3
Bipolar disorder (Psychiatric disorders) | 1 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Cariprazine (3-6 mg/Day) (N=167) | Cariprazine (6-12 mg/Day) (N=169)
Nausea (Gastrointestinal disorders) | 9 | 16 | 19
Constipation (Gastrointestinal disorders) | 5 | 8 | 18
Vomiting (Gastrointestinal disorders) | 10 | 15 | 14
Dyspepsia (Gastrointestinal disorders) | 5 | 7 | 10
Diarrhoea (Gastrointestinal disorders) | 12 | 4 | 9
Akathisia (Nervous system disorders) | 8 | 29 | 38
Headache (Nervous system disorders) | 15 | 19 | 20
Extrapyramidal disorder (Nervous system disorders) | 8 | 16 | 12
Tremor (Nervous system disorders) | 3 | 4 | 10
Dizziness (Nervous system disorders) | 4 | 9 | 7
Insomnia (Psychiatric disorders) | 15 | 16 | 17
Restlessness (Psychiatric disorders) | 8 | 15 | 10

LIMITATIONS AND CAVEATS:
All participants from 1 investigative site were excluded due to Good Clinical Practice (GCP) Violations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.